CLINICAL TRIAL: NCT04159584
Title: Pilot Study: The Effects of Medical Music on Anxiety in Patients With Interstitial Lung Disease
Brief Title: Pilot Study: The Effects of Medical Music on Anxiety in Patients With ILD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Neuralpositive (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1901019911
Record Dates: First submitted 2019-10-22; First posted 2019-11-12 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Intervention Model Description: This is an uncontrolled, interventional pilot study to determine feasibility
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enrolled Subject (Experimental): All subjects will undergo the medical music intervention.
  Interventions: Other: Medical Music

INTERVENTIONS:
Other: Medical Music — Enrolled subjects will undergo 30 minutes of medical music listening

SUMMARY:
This is uncontrolled, interventional feasibility study for determining the effects medical music on anxiety levels in subjects with ILD. Enrolled subjects will be asked to complete questionnaires and undergo physiologic measurements prior to listening to medical music. The music intervention will be for approximately 30 minutes. Post intervention questionnaires and physiologic measurements will be done.

DETAILED DESCRIPTION:
The Medical Music intervention includes playlists that contains songs specifically designed, recorded, and optimized through the provisionally-patented methods, to treat their co-morbid anxiety. The duration of the medical music playlist is 30 minutes.

Enrolled subjects will be asked to complete questionnaires to assess anxiety, a questionnaire related to their music preferences, and undergo physiological measurements (vital signs, galvanic skin response, and heart rate variability) before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 50 to 80 years old
* Diagnosis of definite or probable interstitial lung disease (ILD)
* Willingness to participate and sign consent

Exclusion Criteria:

* Patients who are deaf
* Inability to provide informed consent
* Pregnant women

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of using a medical music intervention as a treatment for anxiety in subjects with ILD, as measured by descriptive evaluation. | Baseline to 30 minutes

SECONDARY OUTCOMES:
Change in State Anxiety Inventory scores before and after intervention | Baseline to 30 min
  The State-Trait Anxiety Inventory Questionnaire is a psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis. It measures two types of anxiety - state anxiety, or anxiety about an event, and trait anxiety, or anxiety level as a personal characteristic.
Change in Visual Analogue Scale scores for Anxiety and Distress (VAS-A) before and after intervention | Baseline to 30 min
  The VAS-A is a psychometric response scale to measure respondents level of anxiety and stress by indicating a position along a continuous line between two end-points ("not at all" to "extremely").
Change in Borg Dyspnea Scale scores before and after intervention | Baseline to 30 min
  The Borg Dyspnea Scale measures perceived dyspnea on a scale from 0 to 10.
Change in heart rate variability before and after intervention | Baseline to 30 min
  Heart rate variability will be measured before and after intervention
Change in galvanic skin response before and after intervention | Baseline to 30 min
  Galvanic skin response will be measured before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kaner, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available to the public upon request in a timely fashion.
Time Frame: 6 months after the publication
Access Criteria: De-identified data will be available to the public upon request in a timely fashion.